CLINICAL TRIAL: NCT01895608
Title: Cognitive Training and Dual-task Ability in Older Adults
Brief Title: Cognitive Training and Dual-task Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E7614-P
Record Dates: First submitted 2013-06-19; First posted 2013-07-10 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-04

CONDITIONS: Gait Disorder
Keywords: aged or aged 80 and over; gait disorder; attention
MeSH Terms: conditions — Mobility Limitation | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Balance rehabilitation + dual-tasking (Experimental): Balance rehabilitation will involve a structured framework of balance activities that require increasing levels of complexity and multimodal stimuli and response demands with the addition of cognitive tasks, (e.g., counting backwards or reciting lists) to be added when the participant can safely perform the primary balance or gait task.
  Interventions: Behavioral: Balance rehabilitation + dual-tasking
- Standard balance rehabilitation (Active Comparator): Standard balance rehabilitation will involve a structured framework of balance activities that require increasing levels of complexity and multimodal stimuli and response demands.
  Interventions: Behavioral: Standard balance rehabilitation
- Cognitive training (speed of processing) (Experimental): Speed of processing cognitive training involves systematically increasing the complexity of visual tasks. Task demands are increased by reducing stimulus duration, adding visual or auditory distractors, increasing number of concurrent tasks or increasing the visual field.
  Interventions: Behavioral: Cognitive training (speed of processing)
- Cognitive training (general cognition) (Active Comparator): General cognitive training involves systematic training of 14 key cognitive abilities, including visual scanning, response time, eye-hand coordination, spatial perception, and working memory. Initial starting point is determined by the software using baseline evaluation.
  Interventions: Behavioral: Cognitive training (general cognition)

INTERVENTIONS:
Behavioral: Balance rehabilitation + dual-tasking — Balance rehabilitation will involve a structured framework of balance activities that require increasing levels of complexity and multimodal stimuli and response demands with the addition of cognitive tasks, (e.g., counting backwards or reciting lists) to be added when the participant
  Arms: Balance rehabilitation + dual-tasking
Behavioral: Standard balance rehabilitation — Standard balance rehabilitation will involve a structured framework of balance activities that require increasing levels of complexity and multimodal stimuli and response demands.
  Arms: Standard balance rehabilitation
Behavioral: Cognitive training (speed of processing) — Speed of processing cognitive training involves systematically increasing the complexity of visual tasks. Task demands are increased by reducing stimulus duration, adding visual or auditory distractors, increasing number of concurrent tasks or increasing the visual field.
  Arms: Cognitive training (speed of processing)
Behavioral: Cognitive training (general cognition) — General cognitive training involves systematic training of 14 key cognitive abilities, including visual scanning, response time, eye-hand coordination, spatial perception, and working memory. Initial starting point is determined by the software using baseline evaluation.
  Arms: Cognitive training (general cognition)

SUMMARY:
The first goal of this study is to examine the extent to which the inclusion of dual-task practice to standard balance rehabilitation results in greater benefits to dual-task ability. The second goal of this study is to examine the extent to which the addition of cognitive training following balance rehabilitation results in greater benefits to dual-task ability.

DETAILED DESCRIPTION:
Historically, degradation of balance control in older adults has been attributed to impairments of the motor and/or sensory systems. As a result, therapy has focused on motor and sensory impairments. However, evidence suggests that an impaired ability to allocate attentional resources to balance during dual-task situations is a powerful predictor of falls. Despite this fact, few studies have examined whether interventions can improve older adults' dual-task ability. The goal of this study is to develop effective interventions to improve ability to allocate attention to balance and gait under dual-task conditions.

Older adults (n = 44) who have been referred to physical therapy (PT) for gait or balance impairments who have dual-task impairment will be randomized to receive either standard balance rehabilitation or balance rehabilitation with dual-task practice. Following PT, subjects will receive cognitive training (CT), either speed of processing or generalized cognitive training. Primary outcomes are ability to walk while performing four different cognitive tasks of varying difficulty. Assessment will occur at baseline, post-PT, post-CT.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include:
* > 60 years of age
* documented balance or mobility problems
* dual-task impairment (timed up and go with subtraction task > 15 s)

Exclusion Criteria:

* Exclusion criteria include:
* cognitive impairment (> 2 errors on Short Portable Mental Status Questionnaire41)
* progressive medical issues that would impact mobility (e.g., Parkinson's disease).

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Hall, PhD PT, Principal Investigator — Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN, Mountain Home, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Balance Rehabilitation + Dual-task Practice: Balance rehabilitation will involve a structured framework of balance activities that require increasing levels of complexity and multimodal stimuli and response demands with the addition of cognitive tasks, (e.g., counting backwards or reciting lists) to be added when the participant can safely perform the primary balance or gait task.
  Balance rehabilitation + dual-task practice: Balance rehabilitation will involve a structured framework of balance activities that require increasing levels of complexity and multimodal stimuli and response demands with the addition of cognitive tasks, (e.g., counting backwards or reciting lists) to be added when the participant
Period: Overall Study
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Started | 10 | 7 | 11 | 6
Completed | 10 | 6 | 8 | 6
Not Completed | 0 | 1 | 3 | 0
Not completed — change in health status | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition) | Total
Number analyzed (Participants) | 10 | 7 | 11 | 6 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.0 (8.3) | 81.9 (7.9) | 78.1 (6.7) | 80.7 (11.1) | 79.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 5 | 3 | 16
  Male | 2 | 7 | 6 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 7 | 11 | 6 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 8 | 6 | 9 | 5 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 11 | 6 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change Scores in Timed up and go With Cognitive Task
Description: Timed up and go test (TUG) has three conditions: no secondary task (TUG), cognitive (TUGc) and manual dual-tasks (TUG-m). Time to complete the task with the cognitive task was recorded as a primary outcome measure. Time greater than 15 s for TUG-c indicates impaired dual-task ability.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Number analyzed (Participants) | 10 | 6 | 8 | 6
seconds | -0.89 (3.36) | -0.37 (2.24) | -0.64 (1.62) | -1.42 (1.92)
Statistical Analysis 1: Comparison: Balance Rehabilitation + Dual-task Practice vs Standard Balance Rehabilitation; Null hypothesis: There will not be a difference in improvement in walking under dual-task conditions following balance rehabilitation that incorporates dual-task practice compared to standard balance rehabilitation; Test type: Other — non-parametric statistic: Mann-Whitney U test for independent samples; p = 0.562, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cognitive Training (Speed of Processing) vs Cognitive Training (General Cognition); Null hypothesis: There will not be a difference in improvement in walking under dual-task conditions following cognitive training that incorporates speed of processing tasks compared to general cognitive training; Test type: Other; p = 0.414, Wilcoxon (Mann-Whitney); non-parametric statistical analysis: Mann Whitney U Test for independent samples

2. Secondary Outcome: Change Scores in Walk While Talk Test With Verbal Fluency Task
Description: The walk while talk (WWT) test involves walking at preferred speed while performing a verbal fluency task.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Number analyzed (Participants) | 10 | 6 | 8 | 6
seconds | 1.76 (3.48) | -3.83 (9.66) | -2.73 (4.67) | 3.01 (10.04)
Statistical Analysis 1: Comparison: Balance Rehabilitation + Dual-task Practice vs Standard Balance Rehabilitation; [analysis description as in outcome 1, analysis 1]; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.181, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cognitive Training (Speed of Processing) vs Cognitive Training (General Cognition); [analysis description as in outcome 1, analysis 2]; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 1.000, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change Scores in Dynamic Gait Index
Description: Dynamic Gait Index (DGI) assesses gait under 8 conditions and has excellent interrater as well as test-retest reliability.
  Each of the 8 conditions is scored on a scale from 0 (indicating severe impairment) to 3 (indicating normal ability). The total score is used for statistical analysis with a maximum score of 24 and a minimum score of 0 with a higher score indicating better performance. A total DGI score less than 20 out of 24 indicates fall risk.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Number analyzed (Participants) | 10 | 6 | 8 | 6
units on a scale | 2.50 (2.07) | 1.50 (4.64) | -0.38 (1.92) | 0.00 (2.45)
Statistical Analysis 1: Comparison: Balance Rehabilitation + Dual-task Practice vs Standard Balance Rehabilitation; Null hypothesis: There will not be a difference in improvement in fall risk as measured by dynamic gait index following balance rehabilitation that incorporates dual-task practice compared to standard balance rehabilitation; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cognitive Training (Speed of Processing) vs Cognitive Training (General Cognition); Null hypothesis: There will not be a difference in improvement in fall risk as measured by dynamic gait index following cognitive training that incorporates speed of processing tasks compared to general cognitive training; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.662, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change Scores in Sensory Organization Test (SOT)
Description: SOT is organized into a series of 6 conditions of increasing difficulty: 3 involve a firm surface with eyes open, eyes closed and with vision sway-referenced and 3 involve a sway-referenced surface with eyes open, eyes closed, and with vision sway-referenced. SOT has good reliability and differentiates fallers and nonfallers.
  The SOT composite score is used for statistical analysis with a maximum score of 100 (indicating perfect stability) and a minimum score of 0 (indicating severe instability). Higher scores indicate better performance (i.e., greater postural stability) and SOT composite scores less than 38 out of 100 indicate fall risk.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Number analyzed (Participants) | 10 | 6 | 8 | 6
units on a scale | 6.44 (12.03) | -1.50 (5.65) | -0.50 (20.28) | 8.60 (6.19)
Statistical Analysis 1: Comparison: Balance Rehabilitation + Dual-task Practice vs Standard Balance Rehabilitation; Null hypothesis: There will not be a difference in improvement in static balance as measured by sensory organization test following balance rehabilitation that incorporates dual-task practice compared to standard balance rehabilitation; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cognitive Training (Speed of Processing) vs Cognitive Training (General Cognition); Null hypothesis: There will not be a difference in improvement in static balance as measured by sensory organization test following cognitive training that incorporates speed of processing tasks compared to general cognitive training; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.171, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change Scores in Preferred Gait Speed
Description: Subjects walk at their preferred speed and time to walk 6 m is recorded.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Number analyzed (Participants) | 10 | 6 | 8 | 6
meters per second | 0.07 (0.29) | 0.24 (0.40) | 0.05 (0.51) | 0.16 (0.18)
Statistical Analysis 1: Comparison: Balance Rehabilitation + Dual-task Practice vs Standard Balance Rehabilitation; Null hypothesis: There will not be a difference in improvement in gait speed following balance rehabilitation that incorporates dual-task practice compared to standard balance rehabilitation; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.313, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cognitive Training (Speed of Processing) vs Cognitive Training (General Cognition); Null hypothesis: There will not be a difference in improvement in gait speed following cognitive training that incorporates speed of processing tasks compared to general cognitive training; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.852, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change Scores in Activities-specific Balance-related Confidence
Description: Subjects' decreased confidence in a variety of situations will be measured using the Activities-specific Balance Confidence scale which has good test-retest reliability. Sixteen activities are each assessed on a scale ranging from 0 to 100, where higher scores indicate greater confidence in performing the activity. Item scores are averaged to arrive at a final score, where average scores <67% indicate a greater fall risk.
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: overall percentage of confidence
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Number analyzed (Participants) | 10 | 6 | 8 | 6
overall percentage of confidence | 10.70 (14.44) | 3.16 (7.04) | -0.31 (7.88) | -8.59 (13.62)
Statistical Analysis 1: Comparison: Balance Rehabilitation + Dual-task Practice vs Standard Balance Rehabilitation; Null hypothesis: There will not be a difference in improvement in balance confidence following balance rehabilitation that incorporates dual-task practice compared to standard balance rehabilitation; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.263, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cognitive Training (Speed of Processing) vs Cognitive Training (General Cognition); Null hypothesis: There will not be a difference in improvement in balance confidence following cognitive training that incorporates speed of processing tasks compared to general cognitive training; Test type: Other — non-parametric statistical analysis: Mann Whitney U Test for independent samples; p = 0.181, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Balance Rehabilitation + Dual-task Practice | Standard Balance Rehabilitation | Cognitive Training (Speed of Processing) | Cognitive Training (General Cognition)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 1/6 | 0/8 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balance Rehabilitation + Dual-task Practice (N=10) | Standard Balance Rehabilitation (N=6) | Cognitive Training (Speed of Processing) (N=8) | Cognitive Training (General Cognition) (N=6)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant fell during the assessment visit while on a break between tasks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes